CLINICAL TRIAL: NCT06598488
Title: Beetroot Juice: A Natural Boost for Cardiovascular Health in Postmenopausal Women?
Acronym: BEETBOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Ann-Katrin Grotle, Associate Professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 730456; 730456 (Other: Regional Ethics Committee.)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-menopause
Keywords: Beetroot juice

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental): 4 days of nitrate rich beetroot juice ingestion (Beet it)
  Interventions: Dietary Supplement: Beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator): 4 days of nitrate depleted beetroot juice ingestion (Beet it)
  Interventions: Dietary Supplement: Beetroot juice placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Beetroot juice will be consumed 2 times a day for 4 days before testing plus one shot on experimental testing day 1,5 hours before arrival.
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Beetroot juice placebo — Beetroot juice will be consumed 2 times a day for 4 days before testing plus one shot on experimental testing day 1,5 hours before arrival.
  Arms: Nitrate depleted beetroot juice

SUMMARY:
This study aims to explore the effects of short-term beetroot juice (BRJ) supplementation on cardiovascular health in post-menopausal women. The primary focus is to determine whether BRJ, rich in nitrates that increase nitric oxide (NO) bioavailability, can reduce blood pressure at rest and during exercise, as well as improve oxygen uptake during maximal exercise. Given the increased cardiovascular risk in post-menopausal women due to the loss of estrogen's protective effects, this research seeks to provide a novel, non-pharmacological intervention to enhance cardiovascular function during exercise in this population.

DETAILED DESCRIPTION:
This study aims to evaluate the short-term effects of beetroot juice (BRJ) supplementation on blood pressure and oxygen uptake during exercise in post-menopausal women. Post-menopausal women are at increased risk of cardiovascular disease due to the loss of estrogen, which plays a critical role in nitric oxide (NO) production, a key regulator of blood vessel function and blood pressure. BRJ, rich in dietary nitrates, is converted into NO in the body and may offer a natural means to improve cardiovascular health.

The primary objective is to investigate whether short-term BRJ supplementation can reduce resting and exercise blood pressure and enhance oxygen uptake during maximal exercise, compared to a placebo. The study will also explore the relationship between these cardiovascular responses and blood biomarkers, including nitrate/nitrite levels and inflammatory cytokines.

The study design is a randomized, double-blind, placebo-controlled crossover trial. Post-menopausal women will be randomized into either the BRJ or placebo group, consuming BRJ or nitrate-depleted juice for 4 days, followed by a 7-day washout period before switching to the alternate group. Participants will undergo testing to measure blood pressure and oxygen uptake at rest and during exercise at baseline and after each intervention.

This research is novel and clinically significant, as it explores a non-pharmacological approach to mitigate cardiovascular risks in post-menopausal women. By improving cardiovascular function, this study aims to offer a new strategy for addressing age- and menopause-related increases in blood pressure and declines in exercise capacity.

ELIGIBILITY:
Inclusion criteria:

* Females under the age of 65
* Self-reported absence of menstrual cycle for >1 year
* BMI <30 kg/m2.
* Able to walk on a treadmill and cycle on a stationary bike without problems.
* Proficient in Norwegian and able to provide informed consent.

Exclusion criteria:

* Current or recent (last 5 years) regular smoker or user of nicotine products
* Addictions to alcohol or illegal drugs
* Allergy or intolerance (s) to nitrate or BRJ supplement.
* Diagnosed with cardiovascular disease (e.g., previous acute myocardial infarction or stroke, peripheral artery disease, heart failure), renal, or respiratory (e.g., asthma, sleep apnea).
* Regular usage of nitrate supplements, including beetroot juice
* Hormone replacement therapy.
* Uncontrolled high blood pressure (e.g., resting systolic and diastolic blood pressure >160/110 mmHg)
* Problems with very low blood pressure (e.g., severe dizziness upon standing)
* Diagnosed with diabetes (type 1 or type 2).
* Using blood pressure or glucose-lowering medications
* Close family (parents, siblings, children) history of sudden cardiac death at an early age (<55 for men, <65 for women)
* Judgment by a medical provider that exercise poses an undue burden or risk.
* Cognitive or psychiatric impairment
* Lack of proficiency in Norwegian language oral or writing skills that will hamper the ability to participate in the interventions and fill out questionnaires.

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | After 4 days of intervention
Blood pressure reactivity | After 4 days of intervention
Maximal oxygen consumption | After 4 days of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No